CLINICAL TRIAL: NCT03722719
Title: Effects of Voluntary Pre-contraction of the Pelvic Floor Muscles (the Knack) on Female Stress Urinary Incontinence - Randomised Controlled Clinical Trial
Brief Title: The Knack on Female Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Fatima Fitz, Physiotherapist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2018-10-21; First posted 2018-10-29 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Stress; Physical Therapy Modalities
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (the Knack) (Experimental)
  Interventions: Other: the Knack
- Group II (PFMT) (Active Comparator)
  Interventions: Other: PFMT
- Group III (the Knack + PFMT) (Active Comparator)
  Interventions: Other: The Knack + PFMT

INTERVENTIONS:
Other: the Knack — The Knack consists of voluntary PFM contractions before and during activities that increase abdominal pressure. Such contraction elevates the pelvic floor cranially, with consequent closure of the urethra, vagina and rectum, stabilization of the pelvic floor and avoidance of urine leakage.
  Other Names: Voluntary PFM pre-contraction
  Arms: Group I (the Knack)
Other: PFMT — The rationale underlying intensive PFM strength training is that it might develop the structural support of the pelvis by raising the levator plate to a permanent, higher position within the pelvis and promoting PFM and connective tissue hypertrophy and stiffness. These conditions facilitate automatic and more efficacious activation of motor units (neural adaptation), which impedes descent during activities that increase abdominal pressure.
  Arms: Group II (PFMT)
Other: The Knack + PFMT — These participants will perform the exercises described for both the Knack and PFMT groups at the outpatient clinic and at home.
  Arms: Group III (the Knack + PFMT)

SUMMARY:
The aim of the present study is to test the hypothesis that voluntary pelvic floor muscle pre-contraction (the Knack) (alone) can be a treatment for urine leakage during efforts. For this purpose, the following parameters will be analysed and compared amongst 1) the Knack, 2) pelvic floor muscle training and 3) the Knack + pelvic floor muscle training groups: urine leakage as assessed by the pad test, urinary symptoms, muscle function, quality of life, subjective cure, adherence to exercises in the outpatient setting and at home and perceived self-efficacy of pelvic floor muscle exercises.

The study population will comprise women with mild to moderate stress urinary incontinence or mixed urinary incontinente (with predominant stress urinary incontinence) as assessed by means of the one-hour pad test (leakage ≥2 g). Leakage up to 10 grams will be rated mild stress urinary incontinence and of 11 to 50 grams as moderate stress urinary incontinence. The sample will also include women with grade 2 muscle strength (normal contraction with elevation of the anterior vaginal wall) on the two-finger assessment rated according to the Oxford scale.

The primary outcome measure will be the objective cure of urinary incontinence as assessed by means of the one-hour pad test three months after randomization.

Secondary outcome measures: three-day bladder diary, 1 hour pad test, International Consultation on Incontinence Questionnaire - Short Form, Incontinence Quality of Life Questionnaire, Subjective cure of stress urinary incontinence, Self-efficacy/outcome expectation to pelvic floor muscle exercises, Frequency of the outpatient sessions, adherence to home exercises and pelvic floor muscle function, morphometry, strength and vaginal squeeze pressure.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate stress urinary incontinence or mixed urinary incontinence (with predominance of stress urinary incontinence) as assessed by means of the one-hour pad test (leakage ≥2 g). Mild stress urinary incontinence will be defined as leakage up to 10 g and moderate stress urinary incontinence as leakage of 11 to 50 g.
* Able to have a gynaecological examination

Exclusion Criteria:

* Symptoms of overactive bladder alone
* Chronic degenerative, uncontrolled metabolic, neurological or psychiatric diseases
* Previous participation in a pelvic floor re-education programe and/or previous pelvic floor surgery or currently receiving other treatment for urinary incontinence
* Pelvic organ prolapse greater than stage II according to the Pelvic Organ Prolapse Quantification (POP-Q) system.
* Use of medication for urinary incontinence or medication that interferes with the musculoskeletal system
* Loss of stools or mucus
* Active urinary or vaginal infection in the past three months
* Body mass index ≥35 Kg/m2

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
One-hour pad test | The primary outcome measure will be the objective cure of urinary incontinence as assessed by means of the one-hour pad test three months after randomization.
  The objective cure of urine loss after intervention will be defined as leakage <2 grams.

SECONDARY OUTCOMES:
Three-day bladder diary | Three and six after months after randomization.
  This validated instrument assesses daytime/night-time urine leakage episodes during three consecutive days.
One-hour pad test. | Three and six after months after randomization.
  This test assesses urine leakage (in grams) in situations involving effort.
International Consultation on Incontinence Questionnaire - Short Form. | Three and six after months after randomization.
  A four-item questionnaire that evaluates the impact of symptoms of incontinence on quality of life and outcome of treatment (0-21 overall score, with greater values indicating increased severity).
Incontinence Quality of Life Questionnaire. | Three and six after months after randomization.
  The impact of stress urinary incontinence on quality of life will be assessed by the Incontinence Quality-of-Life Questionnaire. The Incontinence Quality-of-Life Questionnaire evaluates the limitations on human behaviour, psychosocial impact and social embarrassment. The score ranges from 0 to 100 points, and the lower the score, the greater the impact of urinary incontinence on the patient's quality of life.
Subjective cure of stress urinary incontinence. | Three and six after months after randomization.
  The subjective cure will be measured by asking the patients if they were "satisfied" or "dissatisfied" about their condition (urinary incontinence) after treatment. The investigators considered them to be "satisfied" when the patient was happy with the results and did not want a different treatment and "dissatisfied" if the patient desired a treatment other than the initial one.
Frequency of the outpatient sessions | After three and six months of treatment.
  The number of completed exercise sets will be obtained using an exercise diary, and it will be recorded as the mean of the exercise sets per month performed during the three-month therapy intervention for both groups and the number of home exercise sets in both groups will also be assessed at the six-month follow-up.
Self-efficacy/outcome expectation to pelvic floor muscle exercises | Three and six after months after randomization.
  The scale contains 17 questions in the format of a visual analogue scale with answers ranging from 0 (not confident at all) to 100 (the most confident). Thirteen items refer to self-efficacy and four to outcome expectations. The final scores will be obtained by calculating the mean of the items, ranging from 0 to 100, in which higher values are equivalent to more beneficial self-efficacy/outcome expectation to pelvic floor muscle exercises.
Pelvic floor muscle function | After three and six months of treatment.
  Pelvic floor muscle function - assessed through two-finger vaginal palpation. The muscular performance will be graded for Oxford grade scale in 4 levels (0-3): Degree 0 - absent contraction; and Grade 3 - Strong contraction.
Pelvic floor muscle morphometry | After three and six months of treatment.
  The following measurements will be performed: bladder neck mobility, hiatal area, constriction of the levator hiatus (anteroposterior and transverse lengths of hiatus) and pubovisceral muscle thickness.
Pelvic floor muscle strength | After three and six months of treatment.
  The vaginal dynamometer will measure resistance to unidirectional and anteroposterior compression in kilograms/force (kgf). The participants will be requested to perform three maximum voluntary contractions. The best of the three will be registered.
Vaginal squeeze pressure | After three and six months of treatment.
  Vaginal balloon catheter will be used to assess the vaginal squeeze pressure (in cmH20). The best of three consecutive attempts will be registered as the maximum voluntary contractions.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fitz FF, Gimenez MM, de Azevedo Ferreira L, Matias MMP, Bortolini MAT, Castro RA. Effects of voluntary pre-contraction of the pelvic floor muscles (the Knack) on female stress urinary incontinence-a study protocol for a RCT. Trials. 2021 Jul 23;22(1):484. doi: 10.1186/s13063-021-05440-0. PMID 34301324